CLINICAL TRIAL: NCT05832125
Title: Observatory for Patients Treated for Relapsed or Refractory T-cell Acute Lymphoblastic Leukemia With Oncogenetic Features.
Brief Title: Registry of Relapsed/Refractory T-cell Acute Lymphoblastic Leukemia
Acronym: ALLTARGETOBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Aurélie Cabannes-Hamy, Principal Investigator, Versailles Hospital
Other Study IDs: P21/01_ALL TARGET OBS
Record Dates: First submitted 2023-03-13; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Relapsed/Refractory Acute Lymphoblastic Leukemia; T-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to improve the outcome of relapsed and/or refractory T-cell precursor acute lymphoblastic leukemia (T-ALL) patients, and to facilitate the use of oncogenetic targeted therapies in these patients, we set up an observational cohort, collecting clinical and biological information's from patients with T-ALL in relapse or refractory, as well as the use or not of a targeted therapy. The analysis of the cohort will allow us to evaluate the impact of this therapeutic strategies on the patients' fate, and to facilitate access to innovation and personalized medicine for these patients.

DETAILED DESCRIPTION:
Depending on protocol and leukemia subtype, 5-10% of T-ALL patients are primary refractory, and 30-40% of patients will relapse. A new complete remission is attained in 20-40% of patients, but prolonged disease-free survival is observed in only 10-15% of cases. Nelarabine is approved for R/R T-ALL in second relapses, with a CR rate of 36% in the registration study, and an overall survival of 24% at 1 year and 12% at 3 years.

The biological landscape of T-ALL is well characterized, with the identification of at least 10 key recurrently mutated pathways including transcriptional regulation (91% of cases), cell cycle regulation and tumor suppression (84%), NOTCH1 signaling (79%), epigenetic regulation (68%), PI3K-AKT-mTOR signaling (29%), JAK/STAT signaling (25%), RAS signaling (14%), ribosomal function (13%), ubiquitination (9%) and RNA processing (9%). Furthermore, T-ALL cells are dependent upon BCL-XL and upon BCL-2, especially when the T-ALL blasts bear an ETP phenotype. However, genomic data cannot reliably predict the response of leukemic cells to a given treatment, due to interactions of the different cellular pathways affected in a living leukemic cell. Therefore, the combination of genotypic and phenotypic data may overcome this problem.

In France, patients with relapsed or refractory T-ALL (and also T-cell lymphoblastic lymphomas) are already proposed to undergo a genotypic (oncogenetic characterization) and a phenotypic (drug testing assay) characterization as a standard of care procedure. Based on the results obtained in fresh leukemic cells, a national scientific committee may recommend the used of targeted drugs alone or in combination, in the context of a "off-label" or a "compassionate" use (for example : Temsirolimus + Erwiniase + Venetoclax in PI3K-AKT-mTOR mutated ALL / Tofacitinib + Venetoclax in IL7R-JAK-STAT mutated ALL / 5-azacytidine + Venetocax in hypermethylated ALL / ...).

All patients who undergone this procedure will be proposed to be registered in the ALL-Target registry (ALL-target Observatory). After registration, data related to disease history, disease characterization and disease treatment as well as data describing the patient's condition will be collected.

Some patients may receive conventional chemotherapy as a salvage (conventional cohort), others may receive targeted therapy as a salvage (personalized medicine cohort). The aim of the registry is to evaluate the benefit of each treatment strategy in term of response as a primary end point. Comparison between the two cohorts will be performed after adjustment for confounding factors. Results of subgroups will also be reported using descriptive statistics. Secondary endpoints will include safety of the treatment strategy, survival, disease free survival and progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients with relapsed or refractory T-cell precursor ALL or T-cell lymphoblastic lymphoma
* Oncogenetic analysis performed at diagnosis and/or relapse in the central laboratory

Exclusion Criteria:

* Patient who refuse to be registered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older, with relapsed or refractory T cell precursor-ALL or T-cell Lymphoblastic lymphoma, with oncogenetic analysis performed at diagnosis and/or relapse in the central laboratory.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Response rate defined as complete remission and remission without complete hematological recovery (CR + CRi). | 3 months
  Response rate defined as complete remission and remission without complete hematological recovery (CR + CRi).

SECONDARY OUTCOMES:
Performance Status of patients | 3 months
  Eastern Cooperative Oncology Group (ECOG) - Performans Status Scale PS 0 : Fully active, able to carry on all pre-disease performance without restriction PS 4: Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
Biological description of T-ALL | 3 months
  Phenotypic and oncogenetic characterization with mutated signaling pathways
Description of the treatments received | 3 months
  Number and type of treatment lines received, including current treatment
Description of Overall response rate to treatment | 2 years
  Overall response rate defined by partial response rate + complete response rate
Description of the relapse rate | 2 years
  Event of relapse
Description of survival rate | 2 years
  Death
Duration of response | 2 years
  Response
Description of Adverse Events | 2 years
  Adverse Events

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - CHU Amiens Picardie, Amiens
  - Chu Angers, Angers
  - CH Annecy Genevois, Annecy
  - Centre Hospitalier d'Argenteuil, Argenteuil
  - Centre Hospitalier Montfavet Avignon, Avignon
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Hopital Avicenne, Bobigny
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de CAEN, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - CHU Dijon Bourgogne, Dijon
  - CHU Lille, Lille
  - Chu Limoges, Limoges
  - Hospices Civiles de Lyon, Lyon
  - Grand Hopital de l'Est Francilien, Meaux
  - CHU de Montpellier, Montpellier
  - Centre Hospitalier Emile Muller de Mulhouse, Mulhouse
  - CHU Nancy, Nancy
  - Centre anti-cancer Nice : Antoine Lacassagne, Nice
  - CHU de Nice, Nice
  - CHU Nîmes, Nîmes
  - Hopital Saint-Antoine, Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier de Perpignan, Perpignan
  - CHU de Rennes, Rennes
  - CHU Centre Hospitalier Universitaire de Saint-Étienne - Loire, Saint-Etienne
  - ONCOPOLE, Toulouse
  - Centre Hospitalier de Versailles, Versailles
  - Institut Gustave Roussy, Villejuif